CLINICAL TRIAL: NCT06176326
Title: Program Development Study for Developing Ethical Decision Making and Ethical Sensitivity in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Esra Sezer, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HemsirelikOgrencilerindeEtik
Record Dates: First submitted 2023-11-30; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Ethics education; Nursing students,; Ethics; Education
MeSH Terms: interventions — Nursing

STUDY DESIGN:
Intervention Model Description: One-group Pretest-Posttest Experimental Method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation of the Developed Ethics Education Program (Experimental): The developed education program will be implemented as a 7 week-2 hour session.
  Interventions: Other: Ethics Education Program in Nursing

INTERVENTIONS:
Other: Ethics Education Program in Nursing — In the 7-session training program, each session, lasting 2 hours, presented to students the topic headings determined through the needs analysis of the program development study. This education program consists of sessions on the Introduction to Ethics-Bioethics, Principles of Beneficence and Non-maleficence, Autonomy and Responsibility, Informed Consent and Those Lacking Capacity for Consent, Respect for Human Vulnerability and Individual Integrity, Respect for Private Life and Ensuring Confidentiality, Discrimination, Stigmatization, and Cultural Diversity.

SUMMARY:
The goal of this experimental study is to It is the development, implementation and evaluation of an ethics education program aimed at improving ethical decision making and ethical sensitivity in nursing students. The main questions it aims to answer are:

* Is the training program developed to develop ethical decision-making and ethical sensitivity in nursing students effective on students' ethical decision-making levels?
* Is the training program developed to develop ethical decision making and ethical sensitivity in nursing students effective on students' ethical sensitivity level?

The ındependent variable of the study is the developed education program, and the dependent variable is the students' ethical decision-making and ethical sensitivity levels.

Before the training program is applied to the participants, Ethical Sensitivity Scale Adapted to Nursing Students, Ethical Dilemma Test in Nursing, Preliminary Knowledge Test and Information Forms will be applied. During the implementation of the program, educator diaries and student diaries will be evaluated to evaluate the implementation process. At the end of the program implementation, the program will be evaluated. For evaluation purposes, the Curriculum Evaluation Form will be applied. In addition, Ethical Sensitivity Scale Adapted to Nursing Students and Ethical Dilemma Test in Nursing post-tests will be applied.

DETAILED DESCRIPTION:
The program development study will commence with a needs analysis, employing a democratic approach during the needs analysis process. An analysis of existing documents related to ethical education in nursing will be conducted. Studies on the current status and trends of ethical education in nursing in Turkey and worldwide, expert opinions, and a review of international and national documents will be examined to determine the direction of existing efforts. The Taba-Tyler program development model is planned for use in developing the education program. Based on the data obtained from the needs analysis, the education program will be prepared. Following the preparation of the Ethics Education Program, the population of the study consisting of second-year nursing students will be administered the Adapted Ethical Sensitivity Scale for Nursing Students, Nursing Ethical Dilemma Test, and Information Forms. Students who agree to participate will be informed about the research, and their consent will be obtained.

Thirty-four students who agreed to participate were included in the Nursing Ethics Education Program. They attended a 7-session training program, with each session lasting an average of 2 hours. At the conclusion of this training program, an evaluation of the program was conducted, and the second set of data was collected using the same data collection tools. Following a 1-month follow-up period and a 3-month follow-up period, the Adapted Ethical Sensitivity Scale for Nursing Students and the Nursing Ethical Dilemma Test were administered again to complete continuous measurements.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a nursing undergraduate program
* Not having taken the Ethics in Nursing course as part of the student's academic program
* Willingness to voluntarily participate in the study

Exclusion Criteria:

* Having completed the Ethics in Nursing course as part of the academic program
* Not currently enrolled in a nursing undergraduate program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Change from Total Score of the Ethical Sensitivity Scale Adapted for Nursing Students (ESSNS) | Before the education, immediately after the education, one month after the education, three months after the education
  ESSNS the statement is scored on a scale from 1 point (Strongly disagree) to 7 points (Strongly agree). The total score can range from 30 to 210. A high score indicates high ethical sensitivity, while a low score indicates low ethical sensitivity.
  Change=(Before the education, immediately after the education, one month after the education, three months after the education).
Change from Nursing Ethical Dilemma Test Scale "Practical Thinking" Subscale | Before the education, immediately after the education, one month after the education, three months after the education
  The statement includes a six-item expression that students can consider regarding their approach to the moral dilemma scenario indicated on the scale. Students are expected to choose the most important among these statements and prioritize them according to their importance. Based on the responses given to this section of the test, the aim is to determine the students' level of "Practical Thinking (PD) [Practical Considerations= PC]." The minimum achievable PD score on the test is 6, and the maximum PD score is 36.
  Change=(Before the education, immediately after the education, one month after the education, three months after the education).
Change from Nursing Ethical Dilemma Test Scale "Principle Thinking" Subscale | Before the education, immediately after the education, one month after the education, three months after the education
  Students are presented with a six-item statement reflecting their approach to the moral dilemma scenario indicated on the scale. They are expected to choose the most important among these statements and prioritize them according to their own perceived importance. The purpose of this section of the test is to determine the students' level of "Principled Thinking (PT) [Nursing Principled Thinking= NP]." The minimum achievable PT score on the test is 18, and the maximum is 66, based on the responses given in this section.
  Change=(Before the education, immediately after the education, one month after the education, three months after the education).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa Graduate Education Institute, Istanbul, Avcılar, Turkey (Türkiye)